CLINICAL TRIAL: NCT03569046
Title: General Anesthesia With or Without Local Ear Block in Middle Ear Surgeries; A Randomised, Double-blind Trial
Brief Title: General Anesthesia With or Without Local Ear Block in Middle Ear Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abd-Elazeem Abd-Elhameed Elbakry (Other)
Responsible Party: Sponsor-Investigator, Abd-Elazeem Abd-Elhameed Elbakry, assistant professor of anesthesia, Menoufia University
Organization: Menoufia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2017/12/8/8
Record Dates: First submitted 2018-05-18; First posted 2018-06-26 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Tympanum; Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — Anesthesia, Local; Bupivacaine; Anesthetics, General; Anesthesia, General; Antihypertensive Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The same surgeons performed all the operations to ensure consistency in the estimation of the surgical field. To eliminate the observer bias, the observing anesthetist did not attend the induction of block. Also, the operating surgeon was blinded to the pharmacological treatments, anesthesia and performance of the used techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group l (Active Comparator): ear block by local anaesthetic injection 0.25% bupivacaine. general anesthetic by: midazolam 0.02 mg kg-1 , propofol 2-3 mg kg-1 and lidocaine 0.5 mg kg-1 , fentanyl 2 µg kg-1 , atracurium 0.5 mg kg-1 , isoflurane in 50% oxygen/air. hypotensives for deliberate hypotension by nitroglycerine 0.5-10 μg /kg/min and increments of 0.2 mg propranolol
  Interventions: Drug: local anaesthetic injection; Drug: general anesthetic; Drug: Hypotensives
- Group II (Placebo Comparator): ear block by Normal Saline Flush, 0.9% Injectable Solution . general anesthetic by: midazolam 0.02 mg kg-1 , propofol 2-3 mg kg-1 and lidocaine 0.5 mg kg-1 , fentanyl 2 µg kg-1 , atracurium 0.5 mg kg-1 , isoflurane in 50% oxygen/air. hypotensives for deliberate hypotension by nitroglycerine 0.5-10 μg /kg/min and increments of 0.2 mg propranolol
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution; Drug: general anesthetic; Drug: Hypotensives

INTERVENTIONS:
Drug: local anaesthetic injection — ear block by 0.25% bupivacaine
  Other Names: 0.25% bupivacaine
  Arms: group l
Drug: Normal Saline Flush, 0.9% Injectable Solution — ear block by Normal Saline Flush, 0.9% Injectable Solution
  Other Names: saline ear block
  Arms: Group II
Drug: general anesthetic — general anesthetic by midazolam 0.02 mg kg-1 , propofol 2-3 mg kg-1 and lidocaine 0.5 mg kg-1 , fentanyl 2 μg kg-1 , atracurium 0.5 mg kg-1 , isoflurane in 50% oxygen/air.
  Other Names: general anesthesia
Drug: Hypotensives — hypotensives for deliberate hypotension by nitroglycerine 0.5-10 μg /kg/min and increments of 0.2 mg propranolol
  Other Names: deliberate hypotension

SUMMARY:
Background: Proper selection of anesthetic technique is important in middle ear microsurgery. Controlled hypotension in ear surgery decreases blood loss with improved quality of the surgical field, however, it is associated with resistance to vasodilators and delayed recovery from anesthesia. The use of local anesthetic technique alone in middle ear surgery decreases bleeding and reduces postoperative pain, however, pain on injection, noise, and head-neck position had been reported with the increased risk of patient injuries.

This study aimed to compare the effects of local ear block combined with general anesthesia versus general anesthesia alone, regarding intraoperative hemodynamics, anesthetic consumption, recovery characteristics, postoperative pain, adverse effects and postoperative complications.

DETAILED DESCRIPTION:
Eighty adult patients undergoing middle ear surgery (tympanoplasty with or without mastoidectomy) were enrolled in the study. Patients were randomized into two equal groups (40 patients each). A standardized general anesthetic technique was used in both groups. Group I, received general anesthesia combined with ear block using 10 ml of 0.25% bupivacaine and (Group II), received general anesthesia alone combined with ear block using 10 ml saline. Propofol 2-3 mg /Kg was administered to induce anesthesia, which was maintained using isoflurane. Hemodynamic variables, surgical conditions including the quality of the operative field, intraoperative fentanyl, vasodilators (propranolol and nitroglycerine), isoflurane consumption, recovery time, postoperative pain, total analgesics consumption and postoperative complications were recorded

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II status,
* scheduled for tympanoplasty with or without mastoidectomy

Exclusion Criteria:

* patient refusal,
* known allergy to local anesthetics
* cardiovascular diseases (myocardial infarction, hypertension and valvular heart diseases) --- cerebrovascular diseases (including transient ischemic attacks), renal, hepatic insufficiency or coagulation abnormality.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
mean arterial blood pressure | at arrival to the operating room,1 minute after induction of anesthesia,1 minute after surgical incision,then every 15 minutes till the time of complete surgical wound closure. - postoperative every one hour for 4 hours then every 4 hours for 24 hours
  mean arterial blood pressure in mmHg

SECONDARY OUTCOMES:
heart rate | at arrival to the operating room,1 minute after induction of anesthesia,1 minute after surgical incision,then every 15 minutes till the time of complete surgical wound closure. - postoperative every one hour for 4 hours then every 4 hours for 24 hours
  heart rate in beats /minute
quality of the operative field | every 15 minutes from start of the surgical incision till the time of complete surgical wound closure.
  four-point scale from 0=no bleeding (excellent surgical conditions), 1=minimum bleeding (sporadic suction), 2= diffuse bleeding (repeated suction), and 3=abundant (troublesome) bleeding
recovery time | time from stopping of all anesthetics till the patient had Aldrete's score of 9.
  the time from cessation of all anesthetics until complete recovery using the Aldrete's score
postoperative pain | postoperative: at the time that the patient had Aldrete's score of 9. ,then every 4 hours for 24 hours.
  measured by visual analogue scale (from 0 "no pain" to10 "worst imaginable pain")
total analgesic consumption | in the first 24 hours postoperative
  ketorolac consumption in mg
nitroglycerine consumption | during the operation time
  total nitroglycerine consumption in ug
propranolol consumption | during the operation time
  total propranolol consumption in mg
nausea | in the first 24 hours postoperative
  the number of patients who developed nausea
vomiting | in the first 24 hours postoperative
  the number of patients who developed vomiting
headache | in the first 24 hours postoperative
  the number of patients who developed headache
facial palsy | in the first 24 hours postoperative
  the number of patients who developed facial palsy

CONTACTS AND LOCATIONS:
Overall Officials: Abd-Elazeem A Elbakry, M.D, Study Director — Assistant professor
Locations (1):
- Faculty of Medicine, Cairo, Shebin El-kom, Egypt